CLINICAL TRIAL: NCT01912469
Title: Effects of Traumeel®S Tablets on Exercise Induced Muscle Damage and Muscle Soreness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Dr. med. Frank Christoph Mooren (Other)
Collaborators: Biologische Heilmittel Heel GmbH (Industry); University of Giessen (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Frank Christoph Mooren, Prof. Dr. med. Frank Christoph Mooren, University of Giessen
Organization: University of Giessen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEIR-2; 2009-010898-21 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Exercise-induced Muscle Soreness
Keywords: Muscle; exercise; soreness; Damage; Traumeel
MeSH Terms: conditions — Motor Activity | interventions — Traumeel S

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traumeel (Experimental): Traumeel tablets by mouth the total amount for 72 hours will be 26 tablets
  Interventions: Drug: Traumeel
- Placebo (Placebo Comparator): The Placebo tablets (300 mg lactose monohydrate and 1,5 mg magnesium stearate) by mouth the total amount for 72 hours will be 26 tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Traumeel — oral, Day 1: one tablet every 15 minutes for two hours after the exercise test, 6 hours and 10 hours after the exercise test; Day 2 and 3: two tablets thrice daily; Day 4: two tablets in the morning
  Arms: Traumeel
Drug: Placebo — oral, Day 1: one tablet every 15 minutes for two hours after the exercise test, 6 hours and 10 hours after the exercise test; Day 2 and 3: two tablets thrice daily; Day 4: two tablets in the morning
  Arms: Placebo

SUMMARY:
To investigate and compare the effects of Traumeel®S tablets versus placebo on exercise induced muscle damage and muscle soreness for 72 hours after strenuous eccentric exercise test on downhill treadmill.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male
* Age ≥ 18 and ≤ 40 years
* BMI ≥ 18.5 and < 27,5 kg/m2 (WHO standard for normal range BMI) [48]
* Maximum relative oxygen uptake (VO2max) < 53 ml/kg x min
* General state of good health
* Non-smoker
* Medically approved unrestricted participation in sports as shown by diagnostic performance test conducted on treadmill no longer than 3 months prior to study entry
* Willingness to provide signed informed consent

Exclusion Criteria:

* Regular eccentric exercise training
* Weekly training volume ≥ 6 hours
* Use of dietary supplements (incl. high-dosed vitamins and minerals)
* Chronic immune deficiency
* Current infection
* Heart and/or circulation disorders
* Abnormal findings on exercise ECG
* Musculoskeletal disorders
* Any current clinical condition that requires systemic treatment or might have an impact on study objectives
* Hypersensitivity to botanicals of the Compositae family (e.g. Echinacea)
* Lactose intolerance
* Illicit drug or alcohol abuse
* Participation in another clinical trial within 4 weeks prior to study entry

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in post-exercise two baseline levels up to 72-hours of primary muscle damage marker creatine kinase (CK) | 72 hours
Changes in post-exercise two baseline levels up to 72-hours Short Form McGill Questionnaire total scores and separate VAS pain ratings | 72 hours

SECONDARY OUTCOMES:
Changes in post-exercise two baseline levels up to 72-hours of immunomodulators (35 lab parameters) | 72 hours
Changes in post-exercise two baseline levels up to 72-hours of immune status and activation markers (7 lab parameters) | 72 hours
Changes in post-exercise two baseline levels up to 72-hours of maximum isometric strength (thigh flexors and extensors) | 72 hours
Changes in post-exercise two baseline levels up to 72-hours of muscle marker Lactate Dehydrogenase | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Frank C. Mooren, Prof. Dr., Principal Investigator — Department of Sports Medicine, Institute of Sports Science, University of Giessen
Locations (1):
- Department of Sports Medicine, Institute of Sports Science, University of Giessen, Giessen, Germany

REFERENCES:
- [Derived] Muders K, Pilat C, Deuster V, Frech T, Kruger K, Pons-Kuhnemann J, Mooren FC. Effects of Traumeel (Tr14) on Exercise-Induced Muscle Damage Response in Healthy Subjects: A Double-Blind RCT. Mediators Inflamm. 2016;2016:1693918. doi: 10.1155/2016/1693918. Epub 2016 Jul 5. PMID 27478305